CLINICAL TRIAL: NCT01360281
Title: Neuromuscular Electrical Stimulation and Strength Training in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Gama Filho (Other)
Responsible Party: Thais Varanda Dadalto, Universidade Gama Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE00780312000-10
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Knee Osteoarthritis
Keywords: Quadriceps strength; osteoarthritis rehabilitation; NMES
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ECR (Experimental)
  Interventions: Other: ECR
- Control (No Intervention)
- NMES (Experimental)
  Interventions: Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation
  Arms: NMES
Other: ECR — Resisted exercises
  Arms: ECR

SUMMARY:
The purpose of this study is to compare the efficiency of neuromuscular electrical stimulation and of resisted exercises on increasing quadriceps strength, decreasing pain and on recovering motor function of patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* American College of rheumatology criterion for osteoarthritis diagnosis

Exclusion Criteria:

* Patients that have done knee replacement or are about to do.
* Patients with health conditions that are not compatible with the interventions
* Patients that have done intraarticular corticoid

Min Age: 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Change in Quadriceps strength | Before and after an 8 weeks intervention
Change in Pain | Before and after an 8 weeks intervention
Change in Moving function | Before and after an 8 weeks intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Escola de Fisioterapia da Universidade Gama Filho, Rio de Janeiro, Rio de Janeiro, Brazil